CLINICAL TRIAL: NCT05215405
Title: Intermediate Size Expanded Access Program of Venetoclax (ABT-199) in Combination with Navitoclax (ABT-263) for Pediatric Patients with Relapsed or Refractory Acute Lymphocytic Leukemia (ALL) or Lymphoblastic Lymphoma (LL)
Brief Title: Expanded Access Program of Venetoclax and Navitoclax for Pediatric Patients with Relapsed or Refractory ALL or LL
Status: No longer available | Type: Expanded Access
Sponsor: Kathleen Ludwig (Other)
Responsible Party: Sponsor-Investigator, Kathleen Ludwig, Assistant Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: STU-2021-1222
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Relapsed Childhood ALL; Relapsed Childhood Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax; navitoclax

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered orally once daily (QD), continuously. Each dose of venetoclax should be taken with approximately 240 mL of water within 30 minutes after the completion of a meal, preferably breakfast.
  * Day 1 (200 mg equivalent):
    * Patients 20 < 30 kg will take 70 mg
    * Patients 30 < 35 kg will take120 mg
    * Patients 35 to 45 kg will take 200 mg
  * Day 2 onwards (400 mg equivalent):
    * Patients 20 < 30 kg will take 170 mg
    * Patients 30 < 35 kg will take 250 mg
    * Patients 35 to 45 kg will take 400 mg
  Other Names: ABT-199
Drug: Navitoclax — Navitoclax will be administered orally once daily, starting on day 3 of cycle 1 and then may start on day 1 for subsequent cycles. Navitoclax should be taken at the same time each day approximately 24 hours apart. Dosing will be based on the recommended phase II dosing as per the phase I data and subsequent dose recommendations.
  * Patients 20 < 45 kg will take 25 mg
  * Patients 45 kg or more will take 50 mg
  Other Names: ABT-263

SUMMARY:
The overall goal of this expanded access program is to provide Venetoclax and Navitoclax to patients with acute lymphocytic leukemia (ALL) or lymphoblastic lymphoma (LL) who have exhausted standard treatments.

DETAILED DESCRIPTION:
Acute lymphocytic leukemia (ALL) is a cancer of the immature lymphocytes, a type of white blood cell involved in the body's immune system. People with ALL have lymphocytes that do not mature (lymphoblast). Lymphoblasts replace healthy lymphocytes within the bone marrow and other organs in the lymphatic system.

Lymphoblastic lymphoma (LL) is an aggressive form of non-Hodgkin lymphoma. It is relatively rare, accounting for approximately 2% of all non-Hodgkin lymphomas. In lymphoblastic lymphoma, the abnormal lymphoblasts are present in the lymph nodes or thymus gland, whereas in ALL, the abnormal lymphoblasts are mainly in the blood and bone marrow. Clinically, lymphoblastic lymphoma behaves very similarly to ALL, and the two conditions are often treated with the same regimens.

There have been several recent developments in the treatment of B-ALL, the most common cancer seen in pediatrics. While the cure rate of B-ALL is greater than 90%, children with B-ALL are treated with aggressive chemotherapy regimens that frequently result in long-term toxicities (Oeffinge, Hunger) Furthermore, the patients who experience a relapse have poor outcomes despite treatment with additional chemotherapy often followed by allogeneic stem cell transplant (AlloSCT). The primary predictor of outcome for relapsed B-ALL is the time to relapse; patients who relapse after completing chemotherapy have a cure rate of approximately 50% while those who relapse during treatment have a much lower cure rate of 20-30% (Sun).

Apoptotic pathway targeting therapies, such as navitoclax show promise in the treatment of ALL and LL. Venetoclax +Navitoclax in combination with chemotherapy is well tolerated, with few discontinuations or dose reductions from adverse events (AEs) in patients with relapsed/refractory ALL or LL. The preliminary efficacy of Venetoclax

+Navitoclax was promising in a heavily pretreated population of patients including those with prior SCT or CAR-T, with high rates of Complete response (CR)/complete response with incomplete count recovery (Cri)/complete response with incomplete platelet recovery (CRp), and 10/18 (56%) had undetectable minimal residual disease (MRD). Additional correlative biomarker analyses are ongoing (Pullarkat)

ELIGIBILITY:
Inclusion Criteria:

1. The subject, parent or guardian must voluntarily sign and date an informed consent.
2. Subjects must have relapsed or refractory acute lymphoblastic leukemia (ALL) or relapsed or refractory lymphoblastic lymphoma (LL) and have exhausted available therapies of known benefit for ALL/LL. Refractory is defined as persistent disease after at least 2 courses of chemotherapy.
3. Subjects must be ≥4 years of age
4. Subjects must weight ≥20 kg
5. Subjects must have adequate hepatic function:

   a. ALT and AST ≤5 x ULN and bilirubin ≤1.5 x ULN
6. Subjects must have normal creatinine for age or have a calculated creatinine clearance ≥ 60mL/min/1.73m2
7. Subjects must have adequate performance status:

   1. Subjects ≤ 16 years of age: Lansky ≥ 50,
   2. Subjects > 16 years of age: Karnofsky ≥ 50 or ECOG <3
8. Female subjects of childbearing potential (those who are not postmenopausal for at least 1 year or surgically sterile by bilateral oophorectomy, salpingectomy or hysterectomy) and their male partner must practice as least 1 method of birth control during treatment and through at least 30 days after the last dose of investigational drugs.
9. Male subjects who are sexually active with women of child bearing potential must agree to use condoms during treatment.
10. Female subjects of childbearing potential must have negative results for serum or urine pregnancy test.

Exclusion Criteria:

1. Subjects who have CNS disease with cranial involvement that requires radiation
2. Subjects who are less than 100 days post-transplant, or >100 days post-transplant with active Graft-versus-host disease (GVHD), or are still continuing post-transplant immunosuppressant therapy within 7 days prior to the first dose of investigational drug.
3. Subjects who received any of the following prior to the first dose of investigational drug:

   1. A strong or moderate CYP3A inhibitor or inducer within 7 days
   2. Aspirin within 7 days
4. Subjects who have active, uncontrolled infection
5. Subjects who have not recovered to less than Common Terminology Criteria for Adverse Events (CTCAE) grade 2 from clinically significant adverse effect(s)/toxicity(s) of previous therapy.
6. Subjects with malabsorption syndrome or any other condition that precludes enteral administration.
7. Female subjects who are pregnant or breastfeeding. Male subjects who are considering fathering a child within approximately 30 days or donating sperm during treatment, within approximately 90 days after the last dose of venetoclax/navitoclax.

Min Age: 4 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States